CLINICAL TRIAL: NCT00242385
Title: Single-Dose, Double-Blind, Crossover Study to Evaluate the Pharmacokinetic Comparability of ARALAST Fraction IV-1 Alpha1-Proteinase Inhibitor (ARALAST Fr. IV-1) and ARALAST
Brief Title: Pharmacokinetic Study of ARALAST (Human Alpha1- PI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxter Healthcare, Ltd. (New Zealand), Baxter Healthcare Pty. Ltd. (Australia) (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 460501
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Severe congenital Alpha1-Proteinase Inhibitor (Alpha1-PI) deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

ARMS (2):
- ARALAST Fr. IV-1 (Experimental): 60 mg/kg
  Interventions: Biological: Dose of 60 mg/kg Fraction IV-1 Alpha1-Proteinase Inhibitor
- ARALAST (Active Comparator): 60mg/kg
  Interventions: Biological: Dose of 60 mg/kg alpha1-proteinase inhibitor

INTERVENTIONS:
Biological: Dose of 60 mg/kg Fraction IV-1 Alpha1-Proteinase Inhibitor — Subjects meeting the eligibility criteria were randomized to receive either single dose ARALAST alpha1-proteinase inhibitor 60 mg/kg or single-dose ARALAST alpha1-proteinase inhibitor Fr. IV-1 60 mg/kg at 0.2 mL/kg/min during the first treatment period with crossover to the alternate study product during the second treatment period, with a minimum of 7 days between the two treatment periods.
  Arms: ARALAST Fr. IV-1
Biological: Dose of 60 mg/kg alpha1-proteinase inhibitor — Subjects meeting the eligibility criteria were randomized to receive either single dose ARALAST alpha1-proteinase inhibitor 60 mg/kg or single-dose ARALAST alpha1-proteinase inhibitor Fr. IV-1 60 mg/kg at 0.2 mL/kg/min during the first treatment period with crossover to the alternate study product during the second treatment period, with a minimum of 7 days between the two treatment periods.
  Arms: ARALAST

SUMMARY:
The primary purpose of this study is to characterize the pharmacokinetic profile of intravenous Aralast Fraction (Fr.) IV-1, a sterile, stable, lyophilized preparation of functionally intact human Alpha1- Proteinase Inhibitor (α1-PI). This pharmacokinetic study will be a randomized controlled clinical trial with a cross-over design. Twenty-four subjects will be enrolled into the study. Overall study duration will be approximately 6-8 months.

ELIGIBILITY:
Inclusion Criteria:

* The subject or subject´s legally authorized representative has provided written informed consent
* Subject is 18 years of age or older
* Subject has a documented, endogenous plasma Alpha1-PI level < 8 Micromolar
* Subject is of the genotype Pi*Z/Z, Pi*Z/Null, Pi*Null/Null, Pi*Malton/Z, or others, dependent on the approval by the Sponsor
* If the subject is female or of childbearing potential, the subject has a negative urine test for pregnancy within 7 days prior to first study product administration and agrees to employ adequate birth control measures for the duration of the study
* Laboratory results obtained at the screening visit, meeting the following criteria:

  * Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) <= 2 times the upper limit of normal (ULN)
  * Serum total bilirubin <= 2 times ULN
  * Proteinuria < +2 on dipstick analysis
  * Serum creatinine <= 1.5 times ULN
  * Absolute neutrophil count (ANC) >= 1500 cells/mm3
  * Hemoglobin >= 10.0 g/dL
  * Platelet count >= 10^5/mm3
* If the subject is treated with any respiratory medications, including inhaled bronchodilators and inhaled or oral corticosteroids, the subjects´ medication doses were unchanged for at least 14 days prior to first study product administration
* Nonsmoker for a minimum of 3 months prior to first study product administration

Exclusion Criteria:

* The subject has received any Alpha1-PI augmentation therapy (including Aralast and investigational Alpha1-PIs, by any route including intravenous and inhaled) within 42 days prior to first study product administration
* The subject has received an investigational drug or device within 1 month prior to first study product administration, or the subject is currently receiving an investigational drug
* The subject has a known selective immunoglobulin A (IgA) deficiency (IgA level < 15 mg/dL) and/or antibody to IgA
* The subject has a pulmonary exacerbation or had a pulmonary exacerbation in the past 14 days prior to first study product administration
* The subject is pregnant or lactating, or intends to become pregnant during the course of the study
* The subject has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject safety or compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-12-20 (Actual); Primary Completion 2006-06-05 (Actual); Study Completion 2006-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- Australia (4):
  - Adelaide, South Australia
  - Woodville, South Australia
  - Fitzroy, Victoria
  - Nedlands, Western Australia
- New Zealand (3):
  - Otahuhu, Auckland
  - Christchurch
  - Hamilton

REFERENCES:
- [Derived] Li Z, Franke RM, Morris DN, Yel L. Pharmacokinetics and Biochemical Efficacy of an alpha1-Proteinase Inhibitor (Aralast NP) in alpha1-Antitrypsin Deficiency: a Cross-Product Retrospective Comparability Analysis. Pulm Ther. 2022 Sep;8(3):311-326. doi: 10.1007/s41030-022-00199-4. Epub 2022 Aug 24. PMID 36001294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at seven clinical sites in Australia (4 sites) and New Zealand (3 sites) beginning in December 2005.
Pre-assignment Details: All 25 enrolled subjects were assigned to groups.
Groups:
- ARALAST Fr. IV-1 Then Aralast; ARALAST Then ARALAST Fr. IV-1: Subjects were randomized to receive either single dose ARALAST 60 mg/kg or single-dose ARALAST Fr. IV-1 60 mg/kg at 0.2 mL/kg/min during the first treatment period with crossover to the alternate study product during the second treatment period, with a minimum of 7 days between the two treatment periods.
Period: Period 1
Arm/Group | ARALAST Fr. IV-1 Then Aralast | ARALAST Then ARALAST Fr. IV-1
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0
Period: Period 2
Arm/Group | ARALAST Fr. IV-1 Then Aralast | ARALAST Then ARALAST Fr. IV-1
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects With Severe Congenital α1-PI Deficiency: Subjects were randomized to receive either single dose ARALAST 60 mg/kg or single-dose ARALAST Fr. IV-1 60 mg/kg at 0.2 mL/kg/min during the first treatment period with crossover to the alternate study product during the second treatment period, with a minimum of 7 days between the two treatment periods.
Arm/Group | Subjects With Severe Congenital α1-PI Deficiency
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 59 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 14
  New Zealand | 11

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve/Dose
Description: Area under the plasma alpha1-proteinase inhibitor (α1-PI) concentration versus time curve (AUC) calculated by linear trapezoidal method per dose.
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: All study subjects who received at least 1 dose of study product, and provided data suitable for pharmacokinetic analysis
Measure: Median (Full Range); unit: days*kg/mL
Groups:
- ARALAST Fr. IV-1: Single-dose ARALAST Fr. IV-1 60 mg/kg administered at 0.2 mL/kg/min
- ARALAST: Single dose ARALAST 60 mg/kg administered at 0.2 mL/kg/min
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
days*kg/mL | 0.0822 [0.0750 to 0.094] | 0.0920 [0.0804 to 0.098]
Statistical Analysis 1: Comparison: ARALAST Fr. IV-1 vs ARALAST; Test type: Non-Inferiority or Equivalence — To establish bioequivalence in AUC 0-35d divided by the dose administered with a type I error of 5% the calculated two-sided 90% confidence interval were to be contained completely in the margins of equivalence defined as 80% to 125%; Ratio of Geometric Means = 0.928, 90% CI 2-sided [0.858 to 1.002]

2. Secondary Outcome: Total Area Under the Curve Per Dose
Description: Total area under the α1-PI concentration vs. time curve from pharmacokinetic day 0 to time infinity (AUC 0-infinity) per dose
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: Full Analysis Data Set - all study subjects who received at least 1 dose of study product, and provided data suitable for pharmacokinetic analysis
Measure: Median (Full Range); unit: days*kg/mL
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
days*kg/mL | 0.0825 [0.0750 to 0.095] | 0.0928 [0.0812 to 0.099]
Statistical Analysis 1: Comparison: ARALAST Fr. IV-1 vs ARALAST; Test type: Non-Inferiority or Equivalence — To establish bioequivalence in AUC 0-infinity divided by the dose administered with a type I error of 5% the calculated two-sided 90% confidence interval were to be contained completely in the margins of equivalence defined as 80% to 125%; Ratio of Geometric Means = 0.934, 90% CI 2-sided [0.855 to 1.021]

3. Secondary Outcome: Systemic Clearance (CL)
Description: Computed as dose divided by AUC 0-infinity (AUC 0-infinity was calculated as the sum of AUC from time 0 to the time of last quantifiable concentration plus a tail area correction)
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: mL/day
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
mL/day | 951 [782 to 1115] | 856 [782 to 918]

4. Secondary Outcome: Mean Residence Time (MRT)
Description: Computed as total area under the moment curve (AUMC) divided by total AUC
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
days | 6.8 (3.9) [4.5 to 7.8] | 6.9 (2.8) [5.8 to 7.5]

5. Secondary Outcome: Apparent Volume of Distribution at Steady State
Description: Computed as weight-adjusted CL * MRT
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: mL
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
mL | 5606 [4624 to 6162] | 5405 [4454 to 6703]

6. Secondary Outcome: Terminal Half-life
Description: Computed from the terminal or disposition rate constant obtained from log_e -linear fitting using the least squares deviation to the last five quantifiable concentrations above pre-infusion level.
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
days | 4.1 [3.1 to 5.4] | 4.2 [4.0 to 5.2]

7. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum α1-PI concentration following infusion
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/mL
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
mg/mL | 1.7 [1.4 to 1.8] | 1.7 [1.5 to 1.8]

8. Secondary Outcome: Time to Maximum α1-PI Concentration Post-infusion (Tmax)
Description: Time to reach C-max. Tmax is the number of days from infusion to maximum concentration. Samples drawn at the end of infusion are considered to be time zero.
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
days | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

9. Secondary Outcome: Incremental Recovery
Description: Computed from Cmax (mg/ml) divided by dose per kg body weight (mg/kg).
Time Frame: Pharmacokinetic evaluation: 30 minutes pre-infusion up to 35 days post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: (mg/mL) / (mg/kg)
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
(mg/mL) / (mg/kg) | 0.0259 [0.0234 to 0.028] | 0.0258 [0.0237 to 0.027]

10. Secondary Outcome: Adverse Events (AEs)
Description: Investigators assessed severity of AEs (occurring during or after infusions) based on: MILD: Transient discomfort, does not interfere in a significant manner with participant's normal functioning level; Resolves spontaneously or may require minimal therapeutic intervention MODERATE: AE produces limited impairment of function, can require therapeutic intervention; AE produces no sequelae; SEVERE: AE results in marked impairment of function, can lead to temporary inability to resume usual life pattern; AE produces sequelae, which require prolonged therapeutic intervention
Time Frame: Throughout study period (7 months)
Population: Safety Analysis Data Set - all study subjects who had evidence of receiving at least one dose of study medication regardless of any protocol violation.
Measure: Number; unit: Events
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Number analyzed (Participants) | 25 | 25
Events
  Serious AEs | 0 | 0
  Non-Serious AEs - Mild | 43 | 45
  Non-Serious AEs - Moderate | 16 | 12
  Non-Serious AEs - Severe | 2 | 3

ADVERSE EVENTS:
Time Frame: Throughout the entire study period (7 months)
Groups:
- ARALAST Fr. IV-1: Subjects received a single dose of ARALAST Fr. IV-1 60 mg/kg at 0.2 mL/kg/min
- ARALAST: Subjects received a single dose of ARALAST 60 mg/kg at 0.2 mL/kg/min
Arm/Group | ARALAST Fr. IV-1 | ARALAST
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 23/25 | 19/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARALAST Fr. IV-1 (N=25) | ARALAST (N=25)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vessel puncture site bruise (General disorders) | 3 (3) | 2 (6)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Muscle strain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 1 (3)
Lethargy (Nervous system disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs vary per individual PI, but contain common elements. Baxter requires a review of results communications (e.g., for confidential information) ≥60 days prior to submission or communication. Baxter may request an additional delay of up to 60 days (e.g., to allow for intellectual property protection).